CLINICAL TRIAL: NCT03256994
Title: CIRSE Registry for SIR-Spheres in France (CIRT-FR)
Acronym: CIRT-FR
Status: Completed | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Responsible Party: Sponsor
Other Study IDs: CIRT-FR
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Yttrium-90 loaded SIR-Spheres microspheres — Selective internal radiation therapy (SIRT), also called radioembolisation (RE), with SIR-Spheres microspheres is an endovascular procedure, included within the interventional oncologic technologies to treat primary and secondary liver tumours. Using a microcatheter, a precise dose of resin microspheres is released in the hepatic artery, where they are carried into the arterioles and selectively lodge in the tumour microvasculature. The microspheres are loaded with the radioactive yttrium-90, a high-energy beta-emitting isotope with a half-life of 64.1 hours. SIR-Spheres microspheres are manufactured by Sirtex Medical.
Behavioral: QLQ-C30 with HCC module — In order to measure the palliative aspect of RE with SIR-Spheres microspheres, CIRT-FR will incorporate a quality-of-life questionnaire. CIRT-FR will be using EORTC's QLQ-C30 with HCC Module to measure changes in the quality of life of the patient. The quality-of-life questionnaire will be offered to the patient before the treatment, shortly after the treatment (as soon as possible) and at every follow-up. Filling out the quality-of-life questionnaire is entirely voluntary for the patient

SUMMARY:
Selective Internal Radiation Therapy (SIRT), also known as radioembolisation, is a minimal invasive, endovascular treatment for primary and secondary liver tumours. In France, SIR-Spheres are listed as reimbursable by the national health authorities (Haute Autorité de Santé [HAS]). In order to evaluate the reimbursement after five years, all patients treated with SIR-Spheres will be entered into a registry that collects data on the real-life clinical application of SIRT and reports to the national authorities.

DETAILED DESCRIPTION:
Selective internal radiation therapy (SIRT), also called radioembolisation (RE), with SIR-Spheres microspheres is an endovascular procedure, included within the interventional oncologic technologies to treat primary and secondary liver tumours. Using a microcatheter, a precise dose of resin microspheres is released in the hepatic artery, where they are carried into the arterioles and selectively lodge in the tumour microvasculature. The microspheres are loaded with the radioactive yttrium-90, a high-energy beta-emitting isotope with a half-life of 64.1 hours. Following administration, 94% of the radiation is delivered in 11 days.

In France, SIR-Spheres are listed as reimbursable by the national health authorities (Haute Autorité de Santé [HAS]). In order to evaluate the reimbursement after five years, all patients treated with SIR-Spheres will be entered into a registry that collects data on the real-life clinical application of SIRT and reports to the national authorities.

The goal of the research project is to gain a better understanding of the real-life clinical application of radioembolisation with SIR-Spheres and the impact of the treatment in clinical practice. Secondary objectives will be to assess the observed treatment outcomes of SIRT with SIR-Spheres Y-90 resin microspheres in terms of safety, effectiveness, quality of life, technical considerations and diagnosis and treatment-related considerations.

To better understand the palliative aspect of the treatment, acquisition of the change in quality of life is included by means of EORTC's validated quality of life questionnaire QLQ C30 with accompanying HCC module to measure quality of life in patients with hepatocellular carcinoma.

Besides data collection on the initial treatment, it will be advised to collect follow-up data and quality of life data every three months for a minimum of 24 months after treatment.

CIRT-FR is a post-market, prospective, non-randomized, observational study. Patients are only asked to be enrolled when they are treated with SIR-Spheres microspheres as part of their treatment determined by the treating clinician. In no way will participation of the patient in the registry impact their treatment plan, or influence the quality of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary or secondary liver tumours
* Treatment of liver tumours with SIR-Spheres
* Signed informed consent form

Exclusion Criteria:

- Consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In a general manner and according to the Intent-To-Treat principle, no subject will be excluded from the analysis. The primary and secondary endpoint analysis will include all enrolled subjects in CIRT-FR.
  However, patients who are considered for SIR-Spheres treatment but for whom it was decided that they would not be treated will not be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Description of the clinical context in which SIR-Spheres are applied | Baseline, follow-up every 3 months until 24 months
  Context of systemic therapy; intention of treatment; prior hepatic procedures; post hepatic procedures

SECONDARY OUTCOMES:
Adverse events, treatment complications and laboratory assessments | Follow-up every 3 months until 24 months
  Adverse events measured according to CTCAE 4.03, treatment complications reported bz investigators and abnormal laboratory assessments according to CTCAE 4.03
Effectiveness | Follow-up every 3 months until 24 months
  Based on overall survival (OS), progression free survival (PFS), liver specific PFS
QLQ-C30 | Every 3 months until 24 months
  Quality of life using QLQ-C30 from baseline until 24 months
Technical considerations | Baseline
  Assessed by patient related characteristics, treatment related characteristics, treatment administration and procedure-related outcomes
Diagnosis- and treatment-related considerations | Baseline
  Assessed by type of liver cancer, intention of the treatment, prior hepatic procedures, associated systemic therapy and post-SIRT hepatic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Valérie I Vilgrain, Prof, Study Chair — Cardiovascular and Interventional Radiological Society of Europe; Thomas I Helmberger, Prof, Study Chair — Cardiovascular and Interventional Radiological Society of Europe
Locations (13):
- France (13):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Chu de Dijon, Dijon
  - CHU de Grenoble Alpes, Grenoble
  - Centre Léon Bérard, Lyon
  - CHU de Lyon, Lyon
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nimes, Nîmes
  - Institut Gustave Roussy, Paris
  - CHU de Poitiers, Poitiers
  - CHRU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reimer P, Vilgrain V, Arnold D, Balli T, Golfieri R, Loffroy R, Mosconi C, Ronot M, Sengel C, Schaefer N, Maleux G, Munneke G, Peynircioglu B, Sangro B, Kaufmann N, Urdaniz M, Pereira H, de Jong N, Helmberger T. Factors Impacting Survival After Transarterial Radioembolization in Patients with Unresectable Intrahepatic Cholangiocarcinoma: A Combined Analysis of the Prospective CIRT Studies. Cardiovasc Intervent Radiol. 2024 Mar;47(3):310-324. doi: 10.1007/s00270-023-03657-x. Epub 2024 Feb 6. PMID 38321223
- [Derived] Loffroy R, Ronot M, Greget M, Bouvier A, Mastier C, Sengel C, Tselikas L, Arnold D, Maleux G, Pelage JP, Pellerin O, Peynircioglu B, Sangro B, Schaefer N, Urdaniz M, Kaufmann N, Bilbao JI, Helmberger T, Vilgrain V; CIRT-FR Principal Investigators. Short-term Safety and Quality of Life Outcomes Following Radioembolization in Primary and Secondary Liver Tumours: a Multi-centre Analysis of 200 Patients in France. Cardiovasc Intervent Radiol. 2021 Jan;44(1):36-49. doi: 10.1007/s00270-020-02643-x. Epub 2020 Sep 25. PMID 32975600